CLINICAL TRIAL: NCT02421367
Title: A Phase 1/2, Randomized, Observer-blind Study of Varying Injection Schedules of a Tetravalent Dengue Virus Purified Inactivated Vaccine (TDENV-PIV) With AS03B Adjuvant and Placebo in Healthy Adults in the US
Brief Title: Study of Varying Injection Schedules of TDENV-PIV Vaccine With AS03B Adjuvant and Placebo in Healthy US Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-14-13; WRAIR # 2195 (Other: WRAIR); 201658 (Other: GSK)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TDENV-PIV (0-1) (Experimental): The intervention is a tetravalent dengue virus purified inactivated vaccine (1µg/DENV type) with adjuvant, AS03B.
  The placebo is sodium chloride.
  TDENV-PIV vaccine and placebo will be administered in a single 0.5 mL dose intramuscularly in the non-dominant (whenever possible) deltoid region of the upper arm.
  The intervention will be administered on Day 0 and Day 28. The placebo will be administered on Day 84 and Day 168.
  Interventions: Biological: TDENV-PIV with AS03B adjuvant. Placebo: 0.9% Sodium Chloride Solution.
- TDENV-PIV (0-1-6) (Experimental): The intervention is a tetravalent dengue virus purified inactivated vaccine (1µg/DENV type) with adjuvant, AS03B.
  The placebo is sodium chloride.
  TDENV-PIV vaccine and placebo will be administered in a single 0.5 mL dose intramuscularly in the non-dominant (whenever possible) deltoid region of the upper arm.
  The intervention will be administered on Day 0, Day 28, and Day 168. The placebo will be administered on Day 84.
  Interventions: Biological: TDENV-PIV with AS03B adjuvant. Placebo: 0.9% Sodium Chloride Solution.
- TDENV-PIV (0-3) (Experimental): The intervention is a tetravalent dengue virus purified inactivated vaccine (1µg/DENV type) with adjuvant, AS03B.
  The placebo is sodium chloride.
  TDENV-PIV vaccine and placebo will be administered in a single 0.5 mL dose intramuscularly in the non-dominant (whenever possible) deltoid region of the upper arm.
  The intervention will be administered on Day 84 and Day 168. The placebo will be administered on Day 0 and Day 28.
  Interventions: Biological: TDENV-PIV with AS03B adjuvant. Placebo: 0.9% Sodium Chloride Solution.

INTERVENTIONS:
Biological: TDENV-PIV with AS03B adjuvant. Placebo: 0.9% Sodium Chloride Solution. — Tetravalent dengue virus purified inactivated vaccine (1 µg/virus type)

SUMMARY:
This study is being conducted to evaluate the safety and immunogenicity and antibody persistence of the candidate dengue vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to provide written informed consent.
2. Subjects must be healthy as established by medical history and clinical examination at study entry
3. Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, etc.)
4. Subjects at WRAIR CTC must be able to pass Department of Defense (DoD) base entry requirements, including the possession of a valid government issued ID card.
5. Male or non-pregnant, non-breastfeeding female between 20 and 49 years of age (inclusive) at the time of consent
6. Female subjects of non-childbearing potential (non-childbearing potential is defined as having had one of the following: a tubal ligation at least 3 months prior to enrollment, a hysterectomy, an ovariectomy, or is post-menopausal).
7. Female subjects of childbearing potential may be enrolled in the study, if all of the following apply:

   * Practiced adequate contraception (see Definition of Terms, section 5) for 30 days prior to vaccination
   * Has a negative urine pregnancy test on the day of vaccination
   * Agrees to continue adequate contraception until two months after completion of the vaccination series.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines/placebo during the period starting 30 days preceding the first dose of study vaccine/placebo and/or planned use during the study period
2. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first vaccine/placebo dose (for corticosteroids, this will mean prednisone >=5mg/day or equivalent; inhaled, intranasal and topical steroids are allowed)
3. Planned administration or administration of a vaccine/product not planned in the study protocol during the period starting 30 days prior to the first dose of vaccine/placebo until 30 days after the last dose of study vaccine/placebo (routine influenza vaccination will be allowed as long as it is not administered within 14 days of the vaccine/placebo, and will not lead to study exclusion although it should be reported to the PI)
4. History of dengue infection or dengue illness, or history of flavivirus vaccination (e.g., yellow fever, tick-borne-encephalitis virus [TBEV], Japanese encephalitis, and dengue)
5. Planned administration of any flavivirus vaccine for the entire study duration
6. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device)
7. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required)
8. Family history of congenital or hereditary immunodeficiency
9. Autoimmune disease or history of autoimmune disease
10. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine/placebo or related to a study procedure
11. Major congenital defects or serious chronic illness
12. History of any neurological disorders or seizures
13. Diagnosed with excessive daytime sleepiness (unintended sleep episodes during the day present almost daily for at least 1 month) or narcolepsy; or history of narcolepsy in a subject's parent, sibling, or child
14. Acute disease and/or fever (≥37.5°C/99.5°F oral body temperature) at the time of enrollment: note that a subject with a minor illness such as mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator
15. Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
16. Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the first dose of study vaccine/placebo or planned administration during the study period
17. Recent history of chronic alcohol consumption (more than 2 drinks per day and/or drug abuse (based on subject reported history)
18. Pregnant or breastfeeding female or female currently planning to become pregnant or planning to discontinue adequate contraception
19. A planned move to a location that will prohibit participating in the trial until Study End for the participant
20. Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.
21. Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
22. Safety laboratory test results at screening that are deemed clinically significant or more than Grade 1 deviation from normal

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of solicited local adverse events related to product | 7-day follow-up period after each dose
Intensity of solicited local adverse events related to product | 7-day follow-up period after each dose
Number of unsolicited adverse events related to product | 28-day follow-up period after each dose
Intensity of unsolicited adverse events related to product | 28-day follow-up period after each dose
Number of Grade 2 laboratory abnormalities | 7-day follow-up period after each dose
Number of Grade 3 laboratory abnormalities | 7-day follow-up period after each dose
Number of serious adverse events from day 0 through 28 days after the last dose | 7 months after first dose
Number of potential immune-mediated diseases from Day 0 through 28 days after the last dose | 7 months after first dose
Neutralizing antibody titers to each DENV type | Day 0 and 28 days after the second and third doses of TDENV-PIV
Number of general adverse events related to product | 7-day follow-up period after each dose
Intensity of solicited general adverse events related to product | 7-day follow-up period after each dose
Number of medically attended AEs related to product | Day 0 through 28 days after the last dose

SECONDARY OUTCOMES:
Number of potential immune-mediated diseases from post Month 7 to Study End | 7 months after first dose to the end of study
Number of serious adverse events related to product | 7 months after first dose to the end of study
Neutralizing antibody titers to each DENV type | 56 days after the second dose of active vaccine
Seropositivity status for each DENV type | 28 days after the second dose of active vaccine for all groups
Number of medically attended AEs from post Month 7 to Study End | 7 months after first dose to the end of study
Neutralizing antibody titers to each DENV type for the TDENV-PIV (0-1-6) group | 56 days after the third dose of active vaccine
Neutralizing antibody titers to each DENV type | 4 months after the last dose of active vaccine
Neutralizing antibody titers to each DENV type | 6 months after the last dose of active vaccine
Neutralizing antibody titers to each DENV type | 9 months after the last dose of active vaccine
Neutralizing antibody titers to each DENV type | 12 months after the last dose of active vaccine
Seropositivity status for each DENV type for the TDENV-PIV (0-1-6) group | 28 days after the third dose of active vaccine
Seropositivity status for each DENV type for the TDENV-PIV (0-1-6) group | 56 days after the third dose of active vaccine
Seropositivity status for each DENV type | 4 months after the last dose of active vaccine for all groups
Seropositivity status for each DENV type | 6 months after the last dose of active vaccine for all groups
Seropositivity status for each DENV type | 9 months after the last dose of active vaccine for all groups
Seropositivity status for each DENV type | 12 months after the last dose of active vaccine for all groups

CONTACTS AND LOCATIONS:
Overall Officials: Leyi Lin, M.D., Principal Investigator — USAMRMC/WRAIR
Locations (2):
- United States (2):
  - University of Maryland, Center for Vaccine Development,, Baltimore, Maryland
  - WRAIR, Clinical Trials Center, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin L, Lyke KE, Koren M, Jarman RG, Eckels KH, Lepine E, McArthur MA, Currier JR, Friberg H, Moris P, Keiser PB, De La Barrera R, Vaughn DW, Paris RM, Thomas SJ, Schmidt AC. Safety and Immunogenicity of an AS03B-Adjuvanted Inactivated Tetravalent Dengue Virus Vaccine Administered on Varying Schedules to Healthy U.S. Adults: A Phase 1/2 Randomized Study. Am J Trop Med Hyg. 2020 Jul;103(1):132-141. doi: 10.4269/ajtmh.19-0738. Epub 2020 Apr 23. PMID 32342848